CLINICAL TRIAL: NCT02665130
Title: State Key Laboratory of Respiratory Disease
Brief Title: Comparison of Tai Chi and Pulmonary Rehabilitation on the Effect of Indacaterol in Treatment naïve COPD Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuan-Ming Luo (Other)
Responsible Party: Sponsor-Investigator, Yuan-Ming Luo, State Key Laboratory of Respiratory Disease, State Key Laboratory of Respiratory Disease
Organization: State Key Laboratory of Respiratory Disease (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149BCN01T
Record Dates: First submitted 2015-10-28; First posted 2016-01-27 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tai Ji; indacaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai-Chi group (Active Comparator): Tai-Chi exercise plus Indacaterol 150ug/day
  Interventions: Other: Tai-chi plus Indacaterol
- Pulmonary rehabilitation group (Placebo Comparator): Conventional exercise plus Indacaterol 150ug/day
  Interventions: Other: Pulmonary rehabilitation plus Indacaterol

INTERVENTIONS:
Other: Tai-chi plus Indacaterol — Participants perform Tai-chi exercise 5 days/week and take indacaterol 150ug/day for 24 weeks
  Arms: Tai-Chi group
Other: Pulmonary rehabilitation plus Indacaterol — Participants perform conventional exercise 5 days/week and take indacaterol 150ug/day for 24 weeks
  Arms: Pulmonary rehabilitation group

SUMMARY:
Tai-Chi may be a beneficial form of rehabilitation which is acceptable to the Chinese population but no data exist concerning metabolic responses to Tai-Chi in COPD patients. Investigators conduct an Randomized controlled trial to evaluate the synergistic effect of a Long acting β2-agonists with Tai-Chi as a culturally acceptable form of PR in the Asian population. Classical western style pulmonary rehabilitation will serve as a comparator Investigators propose a prospective randomized controlled trial in which 120 bronchodilator naïve participants (Age 40-80 with GOLD II-IV COPD (post-bronchodilator FEV1 ≥ 25% and <80 % of the predicted normal, and a post-bronchodilator FEV1/FVC < 0.70) are randomized to receive a 26 weeks course of Indacaterol with either Tai-Chi or conventional Pulmonary Rehabilitation. Only participants who are residents in Xingning city (Guangdong Province, China) will be recruited.

Both Tai-Chi and pulmonary rehabilitation will be given by qualified instructors at a rural location in southern China (Xingning). A qualified UK Physiotherapist will also be involved in the management of pulmonary rehabilitation program to further make sure the high quality of pulmonary rehabilitation has been applied. Both arm participants will also receive in an open label fashion Indacaterol 150µg qd. for 6 months giving 2 therapy groups (Tai-Chi/Indacaterol, pulmonary rehabilitation/Indacaterol). The primary endpoint of this study is change in SGRQ between Tai-Chi/Indacaterol and pulmonary rehabilitation/Indacaterol at 14 weeks after entry and the secondary endpoints are change in FEV1% and six minute walk distance. the planned recruitment will be 120 with a view to obtaining 100 completers. The investigators propose the study starts on 31 Dec 2014 and completes on 30 June, 2016.

ELIGIBILITY:
Inclusion Criteria:

1. bronchodilator naïve patients
2. Age 40-80 with GOLD II-IV COPD (post-bronchodilator FEV1 ≥ 25% and <80 % of the predicted normal, and a post-bronchodilator FEV1/FVC < 0.70)
3. patients who are residents in Xingning city (Guangdong Province, China) will be recruited.

Exclusion Criteria:

1. Patients currently or previous on any type of Tai Chi exercise or pulmonary rehabilitation
2. Patients with a history of malignancy of any organ system treated or untreated, within the past 5 years.
3. Patients with clinically significant renal, cardiovascular, neurological, metabolism, immunological, psychiatric, gastrointestinal, hepatic, or haematological abnormalities.
4. Patients with concomitant pulmonary disease (e.g. asthma, lung fibrosis, primary bronchiectasis, sarcoidosis, interstitial lung disorder, tuberculosis)
5. Patients with obesity (BMI> 40 kg/m2).
6. Patients requiring long term oxygen therapy (> 12 h a day) on a daily basis for chronic hypoxemia or recovering from acute exacerbation less than 6 weeks.
7. Patients with Asthma.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
change in St. George's Respiratory Questionnaire (SGRQ) | 14 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Ming Luo, PhD, Principal Investigator — The Affiliated Hospital og Guangzhou Medical University
Locations (1):
- Xing-Ning Hospital, Meizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Polkey MI, Qiu ZH, Zhou L, Zhu MD, Wu YX, Chen YY, Ye SP, He YS, Jiang M, He BT, Mehta B, Zhong NS, Luo YM. Tai Chi and Pulmonary Rehabilitation Compared for Treatment-Naive Patients With COPD: A Randomized Controlled Trial. Chest. 2018 May;153(5):1116-1124. doi: 10.1016/j.chest.2018.01.053. Epub 2018 Apr 3. PMID 29625777